CLINICAL TRIAL: NCT02077543
Title: Molecular and Cellular Print Medical Device Validation in Adult Glioma Tumors
Brief Title: Multicenter Safety Trial Assessing an Innovative Tumor Molecular and Cellular Print Medical Device in Glioma
Acronym: ProTool
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: MEDIMPRINT (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ProTool
Record Dates: First submitted 2013-10-10; First posted 2014-03-04 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Glioma : Oligodendroglioma or Astrocytoma
MeSH Terms: conditions — Astrocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ProTool (Experimental): Device: Brain Tissue Imprint - Medical Device (ProTool)
  Interventions: Device: Brain Tissue Imprint - Medical Device (ProTool)

INTERVENTIONS:
Device: Brain Tissue Imprint - Medical Device (ProTool) — genomic, transcriptomic and proteomic studies.

SUMMARY:
The purpose of the study is to determine the clinical safety and operability of the innovative tissue imprint device ProTool.

DETAILED DESCRIPTION:
Current limitations in the management of high grade brain tumors partly reside in the lack of access to pathological tissue.

Conventional biopsy devices can cause severe side effects, thus limiting the amount of tissue that can be collected for molecular characterization. The Brain-Tissue-Imprint Devices evaluated in this trial offers a unique opportunity to perform multiple non-lesion sampling in both tumor tissue and peritumoral areas. The approach relies on the use of tailored silicon chips integrated in surgical devices enabling tissue sampling through a brief "silicon to tissue contact", thus limiting potential side effects, and opening a way to extensive molecular investigation of brain tumors and their microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old
* patient affiliated to social security or similarly regime
* informed consent form signed
* glial tumor suspicion
* Stereotaxic biopsy indication
* Karnofsky score > 70%
* Hematological assessment :
* neutrophils > 1500/mm3
* Platelet > 150 000
* blood Creatinin normal
* alkaline Phosphatases and transaminases no more than two times normal
* Bilirubin < 1.5 times normal

Exclusion Criteria:

* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Person participating in another clinical study
* Intratumoral hemorrhage MRI detected
* Treatment anticoagulant or antisludge treatments
* Active Infections and non controled or medical affection or psychiatric intercurrent non treated
* Evolutive cerebral oedema without corticoid response
* Non controled Epilepsy without antiepileptics response
* Susceptibility to Medical Device materials allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-10; Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Clinical examination : neurologic deficiency, allergic reaction, infections, pain, headaches, others adverse events... Postoperative MRI evaluation : no hematoma | 2 hours after surgery
Clinical examination : neurologic deficiency, allergic reaction, infections, pain, headaches, others adverse events... Postoperative MRI evaluation : no hematoma | one month after surgery
Clinical examination : neurologic deficiency, allergic reaction, infections, pain, headaches, others adverse events... Postoperative MRI evaluation : no hematoma | 3 months after surgery

SECONDARY OUTCOMES:
Molecular measurements in intra-operative cellular samples : transcriptome, micro-RNA, proteome and cellular cultur analysis | up to 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: François BERGER, MD, PhD, Principal Investigator — University Grenoble Hospital
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Henri Mondor University Hospital, Créteil
  - CLINATEC, Grenoble
  - Grenoble University Hospital, Grenoble
  - Sainte-Anne Hospital, Paris